CLINICAL TRIAL: NCT02143154
Title: Intrapartum Vancomycin in GBS-positive Women: The Effect on Vaginal Group B Streptococcus Colony Counts
Brief Title: Intrapartum Vancomycin for Group B Streptococcus (GBS) Prophylaxis
Status: Completed | Type: Observational
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Other Study IDs: Vancomycin for Group B Strept
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: GBS Positive; Women in Labor Given Vancomycin for Prophylaxis
Keywords: vancomycin, GBS
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — vaginal swabs collected during labor plated for GGBS bacteria and then discarded
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GBS positive women: Women wih GBS positive bacteruria with plan for treatment with vancomycin in labor, or women with positive GBS screening cultures with a plan to receive vancomycin in labor

SUMMARY:
While it is clear that intrapartum antibiotics reduce neonatal GBS infection rates, the mechanism by which these drugs prevent neonatal GBS is not well established. One postulated theory is antibiotics work to reduce bacterial load in the birth canal; thus decreasing fetal exposure during labor and delivery. To our knowledge, the relationship between vancomycin and vaginal GBS colony counts has never been studied. In this prospective cohort study, our objective is to determine the relationship between intrapartum IV vancomycin and vaginal GBS colony counts.

DETAILED DESCRIPTION:
Charts of patients presenting for induction of labor will be reviewed for potential eligibility. After provider permission, eligible patients will be approached for screening who are presenting for induction with documented GBS positivity and plan for vancomycin for intrapartum antibiotic prophylaxis. Patients presenting to the emergency room for labor evaluation/labor evaluation/pre-term labor evaluation, may be pre-screened for potential eligibility. Patients subsequently admitted in labor/preterm labor or with rupture of membranes with documented GBS positivity and plan for vancomycin for intrapartum antibiotic prophylaxis will be approached for screening. Additionally pharmacy will alert study staff when a patient is admitted to the labor floor or antenatal care unit and vancomycin has been ordered for antibiotic prophylaxis. These patients will then be approached for screening

Data collection: Demographic information such as age, race, date of initial GBS culture and time of rupture of membranes will be abstracted from enrolled patients' charts. Intrapartum vaginal cultures will be collected with a vaginal swab from the distal vagina by trained obstetrics and gynecology residents, attendings, nurses, nurse midwives and nurse practitioners prior to the initiation of antibiotics and at two hour intervals until delivery or after eight hours has elapsed.

Swabs will be transported to the lab. Colony counts will be determined via serial dilution. Specimens will be diluted in sterile saline and inoculated onto Columbia Agar containing 5% sheep blood, colistin (10 mg), and nalidixic acid (10 mg/L). After incubation for 48 hours at 35 C in ambient air, the number of colonies on the dilution plates will be visually counted and multiplied by the appropriate dilution factor for that particular plate.

ELIGIBILITY:
Inclusion Criteria:

* Women with documented GBS-positive antenatal screening culture or documented GBS bacteruria during pregnancy with plan to receive vancomycin for intrapartum antibiotic prophylaxis,
* ability to give informed consent,
* aged 18-48,
* English and or Spanish speaking, admitted in labor or undergoing induction of labor

Exclusion Criteria:

* Inability to give consent,
* currently receiving antibiotics for another indication,
* recent antibiotic use (within the previous 7 days),
* allergy to vancomycin

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with documented GBS-positive antenatal screening culture or documented GBS bacteruria during pregnancy with plan to receive vancomycin for intrapartum antibiotic prophylaxis
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2014-10; Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Percentage decline in vaginal GBS colony counts | up to eight hours or delivery

CONTACTS AND LOCATIONS:
Overall Officials: Maureen S Hamel, MD, Principal Investigator — Warren Alpert Medical School of Brown University, Women & Infants Hospital of Rhode Island, Department of Obstetrics and Gynecology
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided